CLINICAL TRIAL: NCT02687087
Title: Assessing the Safety and Effectiveness of Visco-ease for the Treatment of Radiotherapy Induced Xerostomia in Head and Neck Cancer Patients
Brief Title: A Study of Patients With Dry Mouth and Sticky Saliva During Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Lamellar Biomedical Ltd (Industry); University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GN14ON413; 00908 (Other: Funder); 44528835 (Registry Identifier: ISRCTN Registry)
Record Dates: First submitted 2016-02-17; First posted 2016-02-22 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Xerostomia
Keywords: Radiotherapy Induced Xerostomia (RIX)
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visco-ease (Experimental): Visco-ease is a suspension of multilamellar vesicles comprising lipids in ratios which mimic the lipidic composition of endogenous extra-alveolar lamellar bodies. Visco-ease is suspended in physiological saline (0.9% NaCl) to provide a final dose concentration of 19.6 mg/mL. Visco-ease is a white to off-white turbid suspension. The device under evaluation in this clinical investigation is Visco-ease at a concentration of 19.6 mg/mL.
  Interventions: Device: Visco-ease
- RIX-Placebo (Placebo Comparator): Physiological Saline (sodium chloride 0.9% (w/v)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Visco-ease — 19.6 mg/mL of LMS-611
  Other Names: RIX - LMS-611x-20; OXB/1-20; LMS-611
  Arms: Visco-ease
Device: Placebo — Physiological Saline
  Other Names: 0.9% (w/v) Physiological Saline
  Arms: RIX-Placebo

SUMMARY:
The purpose of this study is to evaluate the clinical safety and effectiveness of Visco-ease dry mouth spray for the treatment of Radiotherapy Induced Xerostomia (RIX) in head and neck cancer patients.

A parallel group double blind study design has been selected. The primary outcome is change in GRIX scores from baseline (visit 1) to end of treatment (visit 7). The primary outcome will be compared between Visco-ease and the placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent
2. Male or female subjects ≥ 18 years of age
3. Subjects prescribed radiotherapy or chemoradiotherapy as primary treatment for head and neck tumours where one or more parotid glands will receive a significant dose of radiation as judged by the CI or PI during the radiotherapy planning process

Exclusion Criteria:

1. Subject is pregnant or breastfeeding
2. Subjects with known allergies to egg, soya, or lanolin (sheep's wool grease) based products
3. Subjects with a history of an autoimmune disease with pre-treatment xerostomia (e.g. Sjögren's syndrome) or other underlying systemic illness known to cause xerostomia independent of prior radiation therapy exposure
4. Subjects who have participated in an investigational medicinal product study within 30 days prior to signing consent
5. Any clinically significant disease or condition that may interfere with the study treatment or outcome of the study (at the discretion of the CI or PI)
6. Subjects who are unable to independently complete the questionnaire or diary
7. Subjects who are judged inappropriate for inclusion in the study by the CI or PI
8. Subjects with head and neck cancer who have had surgery to the primary site. Neck dissection alone is not an exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Change in GRIX Score | From baseline (Visit 1) to end of treatment (Visit 7, after 6 weeks of treatment)
  The primary endpoint will compare change in GRIX scores from baseline to 6-week follow-up between the group treated with Visco-ease and the Placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Paterson, Principal Investigator — Beatson West of Scotland Cancer Centre
Locations (1):
- Beatson West of Scotland Cancer Centre, Glasgow, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No